CLINICAL TRIAL: NCT04984720
Title: Efficacy of Smartphone Based Digital Application to Track Migraine, Offer Pill Reminders and Community Blog in Improving Headache Related Parameters as Compared to Paper Pen Diary in Patients With Migraine - Cross Over RCT
Brief Title: Efficacy of Smartphone Based Digital Application in Improving Headache Related Parameters in Patients With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Assistant Professor, Department of Neurology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IECPG-299/28.04.2021
Record Dates: First submitted 2021-07-18; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Migraine
Keywords: Mobile phone application; Behavioural intervention; Headache outcomes; Medication adherence; Quality of life
MeSH Terms: conditions — Migraine Disorders; Medication Adherence

STUDY DESIGN:
Intervention Model Description: * A run-in period of 4 weeks prior to randomization to optimize therapy and to document the baseline frequency and severity of headaches.
  * At the end of run-in period, the patients will be randomly allocated into the smartphone based digital App first arm or the paper diary first arm. The digital app and paper diary- are available in Hindi as well as English.
  * Randomization will be done by computer generated random number table.
  * Concealment: The sequence of allocation will be held concealed by opaque sealed envelopes.
  * Participant and investigator both will be aware of the allocated group - it is an open label study.
  * Participants will be followed up at 4 weeks and the headache characteristics and outcome parameters would be captured from the app and paper diary respectively.
  * Subsequently patients would be crossed over to the other arm and 4 weeks after the cross over, parameters would again be assessed.
Who Masked: Outcomes Assessor
Masking Description: The participant, investigator and care provider will be aware of the intervention and the sequence in which it is administered.
  The outcomes will be assessed by an outcome assessor who will not be aware of the arm into which the participant was randomized prior to the assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart phone based digital app arm (Experimental): Digital smartphone application which tracks migraine and to offers pill reminders for medication adherence and community blog and disease related educational material for migraineurs will be given to the patients
  Interventions: Behavioral: Smartphone based digital application
- Paper and pen diary arm (Active Comparator): Clinic based education and traditional paper-pen diary will be administered in tracking headache parameters
  Interventions: Behavioral: Smartphone based digital application

INTERVENTIONS:
Behavioral: Smartphone based digital application — Smartphone Based Digital Application to Track Migraine, Offer Pill Reminders for Medication Adherence and Community Blog
  Other Names: Paper pen diary

SUMMARY:
Migraine is a common headache disorder and affects 1 in 5 adults during their lifetime. It is a disorder which leads to significantly impaired quality of life, absence from work, loss of productivity in workplace and reduced vitality in social functioning. One of the important cornerstones in the management of migraine is the maintenance of a good headache diary. A headache diary enables the physician to understand the headache characteristics as well to establish the triggers causing the precipitation of episodes. The other important measure to ensure good outcomes is compliance to medications in those who have been prescribed prophylaxis. Migraine prophylaxis is by pills that have to be taken everyday at fixed time to ensure best outcomes. However, it is known that patients with migraine often are not adherent to prophylactic medications. A meta-analysis of 33 studies found that observational studies (n = 14) showed adherence ranging from 41% to 95% at 2 months after initiation of medication and 21% to 80% at 6 months. Pooled rates of persistence derived from 19 RCTs on propranolol, amitriptyline, and topiramate showed adherence rates of 77%, 55%, and 57%, respectively, at 16-26 weeks of initiation. The real world adherence is expected to be lower than that in the ideal settings of randomized trials. Regular pill reminders issued through smartphone based applications can improve medication adherence and thus improve headache outcomes. Though smartphone based migraine tracker digital applications are available, they mostly are aimed at capturing headache characteristics. The efficacy of providing pill reminders along with patient educational materials and community blog to enable migraineurs share their experiences with each other has not been studied in controlled trials. It is known that patients who are well informed about their chronic diseases such as migraine often have better outcomes. Busy clinicians often resort to providing pamphlets regarding the disease, triggers, acute pain relief medications, prophylactic therapy etc. However, it is yet to be studied if a digital application with all these inbuilt features, which are easily accessible at the finger tips would lead to better information uptake and improved compliance and self management. This RCT would try to assess this gap in knowledge.

DETAILED DESCRIPTION:
Migraine is a common headache disorder which leads to significantly impaired quality of life, absence from work, loss of productivity in workplace and reduced vitality in social functioning. A structured migraine diary can be a valuable aid for improving communication between patients and physicians regarding migraine disability and treatment outcomes. The other possible measure to ensure improved outcome in migraine patients is better adherence to prophylactic treatment of migraine. Migraine prophylaxis is by pills that have to be taken every day at fixed time to ensure best outcomes. However, it is known that patients with migraine often are not adherent to prophylactic medications. Regular pill reminders issued through smartphone based applications may help improve medication adherence and hence, headache outcomes. Though smartphone based migraine tracker digital applications are available, they mostly are aimed at capturing headache characteristics. The efficacy of providing pill reminders along with patient educational materials and community blog to enable migraineurs share their experiences with each other has not been studied in controlled trials. It is known that patients who are well informed about their chronic diseases such as migraine often have better outcomes. Busy clinicians often resort to providing pamphlets regarding the disease, triggers, acute pain relief medications, prophylactic therapy etc. However, it is yet to be studied if a digital application with all these inbuilt features, which are easily accessible at the finger tips would lead to better information uptake and improved compliance and self management. This RCT would try to assess this gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients attending neurology OPD.
* At least 18 years of age; any gender.
* Episodic or chronic migraine diagnosed (using International Classification of Headache Disorders-3 (ICHD-3) .
* No modifications to the prophylactic therapy or acute pain relief medications is planned over the next 3 months.
* Can read and write in Hindi or English easily.
* Have an Android/iOS smart phone in which digital application can be installed and who knows how to operate smart phone.
* Ready to provide consent and willing to adhere to protocol and comply with follow up visits.
* No major neurological or systemic medical condition that reduces life expectancy to less than 1 year based on clinical prediction scores.

Exclusion Criteria:

* Not willing to adhere to protocol.
* Not willing to provide consent.
* Inability or unwillingness to complete diary recording.
* Patients with Medication over use headache ( as per ICHD -3).
* Other primary headaches and secondary headache disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-07-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in HIT-6 (Headache impact test-6) score | 4 weeks
  To compare the change in HIT-6 (Headache impact test-6 ranges from 36-78 with a higher score indicating greater severity) score from baseline to 4 weeks after introduction of the digital smartphone based application vs paper-pen diary.
Reduction in headache days | 4 weeks
  To compare the percentage of patients reporting 30 % or more reduction in headache days at 4 weeks following introduction of digital smart phone based application vs paper-pen diary .

SECONDARY OUTCOMES:
Compliance | 4 weeks
  The proportion of patients who comply with using the digital smartphone based application vs paper-pen diary.
Number of headache days per 28 days | 4 weeks
  The number of headache days per 28 days following usage of digital smartphone based application vs paper-pen diary.
Change in number of headache days per 28 days from baseline | 4 weeks
  The change from baseline in number of headache days per 28 days following usage of digital smartphone based application vs paper-pen diary .
change from baseline in the number of days with severe headaches per 28 days | 4 weeks
  The change from baseline in the number of days with severe headaches in the preceding 4 weeks as compared with baseline in patients using the digital smartphone based application vs paper-pen diary.
Change from baseline in the duration of headache episodes in the preceding 4 weeks | 4 weeks
  The change from baseline in the duration of headache episodes in the preceding 4 weeks as compared with baseline in patients using the digital smartphone based application vs paper-pen diary
Headache severity on VAS (Visual analogue scale) | 4 weeks
  Headache severity on VAS scale (0-10 with higher score meaning greater pain) in patients using the digital smartphone based application vs paper-pen diary
Change from baseline in severity of headache on VAS scale (Visual analogue scale) | 4 weeks
  Change from baseline in severity of headache on VAS scale (0-10 with higher score meaning greater pain) in patients using the digital smartphone based application vs paper-pen diary
Number of headache episodes needing rescue medication | 4 weeks
  The number of headache episodes needing rescue medication in patients using the digital smartphone based application vs paper-pen diary.
Change from baseline in need for rescue medication | 4 weeks
  Change from baseline in number of headache episodes needing acute pain relief medications in patients using the digital smartphone based application vs paper-pen diary.
Omission rates | 4 weeks
  Omission rates in daily diary entries in patients using the digital smartphone based application vs paper-pen diary.
Triggers | 4 weeks
  Factors that trigger the onset of headaches (like specific foods, sleep deprivation, travel, etc) in patients using the digital smartphone based application vs paper-pen diary.

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, New Delhi, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request from the investigator through our AIIMS Institute ethics committee, the individual participant data will be made available to other researchers
Supporting Information: Study Protocol, CSR
Time Frame: will be available within 6 weeks for as long as suggested by our institute ethics committee
Access Criteria: Request to be made through the Institute ethics committee and would be processed as per Institute rules